CLINICAL TRIAL: NCT02986737
Title: ACURATE Neo™ Aortic Bioprosthesis for Implantation Using the ACURATE TA™ LP Transapical Delivery System in Patients With Severe Aortic Stenosis
Acronym: TALP-FIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014-02
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Aortic Stenosis
Keywords: TAVI; Aortic Stenosis; Transcatether Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Medical device trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACURATE neo™ and ACURATE TA™ LP (Experimental): Patients implanted with ACURATE neo™ Aortic Bioprosthesis and ACURATE TA™ LP Transapical Delivery System
  Interventions: Device: ACURATE neo™ and ACURATE TA™ LP

INTERVENTIONS:
Device: ACURATE neo™ and ACURATE TA™ LP — ACURATE neo™ Aortic Bioprosthesis and ACURATE TA™ LP Transapical Delivery System on patients with severe aortic stenosis where conventional aortic valve replacement (AVR) via open-heart surgery is considered to be high risk

SUMMARY:
Trial of ACURATE neo(TM) Aortic Bioprosthesis for Implantation using the ACURATE TA(TM) LP Transapical Delivery System in Patients with Severe Aortic Stenosis for evaluating the Safety and performance of the study device

DETAILED DESCRIPTION:
This is a single arm, prospective, multicenter non randomised and open trial of the treatment of patients with severe aortic stenosis where conventional aortic valve replacement (AVR) via open heart surgery is considered to be high risk. All patients will be followed up to 5 years after the intervention.

The primary objective is to evaluate the safety and performance of the study device in patients presenting with severe aortic stenosis considered to be high risk for surgery Secondary objective is to evaluate adverse events and study device performance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 75 years of age and older
2. Severe aortic stenosis defined as:

   Mean aortic gradient > 40mmHg or o Peak jet velocity > 4.0m/sor Aortic valve area of < 1.0cm2
3. High risk candidate for conventional AVR defined as:

   STS score ≥ 10 or Multidisciplinary heart team (cardiologist and cardiac surgeon) consensus that patient is not a surgical candidate for conventional AVR due to significant co- morbid conditions unrelated to aortic stenosis
4. NYHA Functional Class > II
5. Multidisciplinary heart team (cardiologist and cardiac surgeon) consensus that the transapical approach is the most suitable TAVI access route
6. Aortic annulus diameter from ≥ 21mm up to ≤ 27mm by CT or TEE
7. Patient willing to participate in the study and provides signed informed consent

Exclusion Criteria:

1. Congenital unicuspid or bicuspid aortic valve
2. Extreme eccentricity of calcification
3. Severe mitral regurgitation (> Grade 2)
4. Pre-existing prosthetic heart valve in any position and / or prosthetic ring
5. LV apex is not accessible via transapical access due to severe chest deformity
6. Previous surgery of the LV using a patch, such as the Dor procedure
7. Presence of apical LV thrombus
8. Calcified pericardium
9. Septal hypertrophy unacceptable for transapical procedure
10. Transesophageal echocardiogram (TEE) is contraindicated
11. ECHO evidence of intracardiac mass, thrombus, or vegetation
12. LVEF < 30% by ECHO
13. Emergency procedure pre-implant including CAD requiring revascularization
14. Any percutaneous intervention, except for balloon valvuloplasty (BAV) within 1 month prior to implant procedure
15. Acute myocardial infarction within 1 month prior to implant procedure
16. Previous TIA or stroke within 3 months prior to implant procedure
17. Active gastrointestinal (GI) bleeding within 3 months prior to implant procedure
18. Scheduled surgical or percutaneous procedure to be performed prior to 30 day visit
19. History of bleeding diathesis or coagulopathy or refusal of blood transfusions
20. Systolic pressure <80mmHg, cardiogenic shock, need for inotropic support or IABP
21. Primary hypertrophic obstructive cardiomyopathy (HOCM)
22. Active infection, endocarditis or pyrexia
23. Hepatic failure (> Child B)
24. Chronic renal dysfunction with serum creatinine > 2.5 mg/dL or renal dialysis
25. Refusal of surgery
26. Severe COPD requiring home oxygen
27. Neurological disease severely affecting ambulation, daily functioning, or dementia
28. Life expectancy < 12 months due to non-cardiac co-morbid conditions
29. Contraindication to study medication, contrast media, or allergy to nitinol
30. Currently participating in an investigational drug or another device study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days
  incidence of all cause mortality at 30 days
Mean aortic gradient after device implantation | 7 days or Discharge
  mean aortic gradient evaluated by echocardiography and by the site at 7days or discharge per standard post-implantation follow-up

SECONDARY OUTCOMES:
rate of clinical endpoints VARC II | 30 days and month 12
  rate of clinical endpoints VARC II at 30 days and 12 months
procedural success | procedure
  procedural success defined as ACURATE neo™ at intended location
device success assessed according to composite VARC 2 criteria | 7 days, 30 days, 12 months
  Device success defined as:
  * ACURATE neo™ implanted in intended location
  * No impingement of the mitral valve
  * Normal coronary blood flow
  * Insufficiency < Grade 3
  * Mean aortic gradient < 20mmHg
  * EOA ≥ 1.0 cm2 No further re-intervention performed on the ACURATE neo™ implant
functional improvement from Baseline as per NYHA Functional Classification | 30 days and 12 months follow up
  functional improvement from baseline as per NYHA functional classification at 30 days and 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mirko Doss, Prof.Dr.Med, Principal Investigator — Abteilung Herzchirurgie Kerckhoff-Klinik
Locations (2):
- Germany (2):
  - Kerckhoff-Klinik, Bad Nauheim
  - Klinik für Herz-und Gefäßchirurgie, Hamburg

IPD SHARING:
Plan to Share IPD: No